CLINICAL TRIAL: NCT03842878
Title: Prospective, Longitudinal Study of the Natural History and Functional Status of Patients With Limb-Girdle Muscular Dystrophy 2I
Brief Title: Natural History Study of Patients With Limb-Girdle Muscular Dystrophy 2I
Status: Completed | Type: Observational
Sponsor: Genethon (Other)
Responsible Party: Sponsor
Other Study IDs: GNT-015-FKRP
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2024-06

CONDITIONS: LGMD2I
MeSH Terms: conditions — Muscular Dystrophy, Limb-Girdle, Type 2I

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, longitudinal, interventional, single-group, multicenter natural history study to better know the LGMD2I disease physiopathology. The duration of participation for each patient will be up to 24 months.

DETAILED DESCRIPTION:
Study duration Duration from First visit of first patient (FPFV) to Last visit of last patient (LPLV) : 3 years

Study objectives Primary objective:

To characterize the disease course in Limb-Girdle Muscular Dystrophy 2I (LGMD2I) patients using standardized and disease appropriate evaluations.

Secondary objectives:

To identify clinical, imaging and/or laboratory parameters that are indicators of the disease course in LGMD2I To identify the best outcome measure for further therapeutics approaches

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients
2. Patients ≥ 16 years old
3. Clinical diagnosis of LGMD2I and gene testing demonstrating two pathogenic mutations in fukutin-related protein gene, FKRP)
4. Ambulant patients

Exclusion Criteria:

1. Patients presenting other disease which may significantly interfere with the interpretation of LGMD2I natural history

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female and male patients ≥ 16 years old
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
6-Minute Walk Test | Baseline through 24 months
  Primary endpoint
10-Meter Walk test (10MWT) | Baseline through 24 months
  Primary endpoint
Timed Up and Go (TUG) test | Baseline through 24 months
  Primary endpoint
Four-stair climb test | Baseline through 24 months
  Primary endpoint
North Star Assessment for Neuromuscular Disorders (NSAD) | Baseline through 24 months
  Scale to assess patient's abilities necessary to remain functionnaly ambulant
Upper limb assessment via the Performance of the Upper Limb (PUL) tool version 2.0 | Baseline through 24 months
  Primary endpoint
Recording of aids for ambulation | Baseline through 24 months
  Primary endpoint
Isokinetic muscle testing using the Biodex System (optional) | Baseline through 24 months
  Primary endpoint
Pulmonary function test | Baseline through 24 months
  Primary endpoint
Electrocardiogram | Baseline through 24 months
  Presence of cardiac abnormalities or any ventricular extrasystoles will be investigated
Echocardiography | Baseline through 24 months
  Cardiac dimensions will be measured to investigate the presence of any dilated cardiomyopathy

CONTACTS AND LOCATIONS:
Overall Officials: John Vissing, PR, Principal Investigator — Professor of neurology
Locations (3):
- Pr John Vissing, Copenhagen, Denmark
- Dr Tanya Stojkovic, Paris, France
- Pr Volker Straub, Newcastle, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided